CLINICAL TRIAL: NCT04589247
Title: Improving Cancer Care by Incorporating the Patient's Voice Into On-treatment Symptom Management
Brief Title: Improving Cancer On-treatment Symptom Management
Acronym: IMPROVE
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: WellSpan Health (Other)
Responsible Party: Sponsor
Other Study IDs: J2048; IRB00218263 (Other: JHM IRB)
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Thoracic Neoplasms; Gastrointestinal Cancer; Lung Cancer
Keywords: Patient Reported Outcomes; Radiotherapy
MeSH Terms: conditions — Neoplasms; Thoracic Neoplasms; Gastrointestinal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer treated with definitive-intent radiotherapy: Histologically confirmed loco-regional to advanced primary cancer, including but not limited to lung cancer, esophageal, or gastro-intestinal cancers at risk of developing radiotherapy-related toxicity.

SUMMARY:
Patient-reported outcome measures (PROMs) is an umbrella term that refers to any report on a health status measure that is reported directly by the patient, without the influence of clinicians or anyone else. PROMs have been shown to more closely reflect a patient's daily health status when compared to physician-reported measures. However, research is needed to evaluate if patient symptom reporting during definitive-intent radiotherapy allows earlier and improved detection of treatment toxicity.

The IMPROVE pilot study will describe the proportion of patients with cancer with changes in physician-perception of treatment-related toxicity that result from routine physician review of PROMs reported during definitive radiotherapy.

DETAILED DESCRIPTION:
Patient-reported outcome measures (PROMs) is an umbrella term that refers to any report on a health status measure that is reported directly by the patient, without the influence of clinicians or anyone else. PROMs have been shown to more closely reflect a patient's daily health status when compared to physician-reported measures. However, research is needed to evaluate if patient symptom reporting during definitive-intent radiotherapy allows earlier and improved detection of treatment toxicity, and leads to individualized interventions which may improve the toxicity outcomes for patients with locally-advanced and oligometastatic cancer.

The investigators hypothesize that routine physician review of PROMs during on-treatment visits will (1) increase proportion of patients with an increased in their physician' s assessment of their overall toxicity burden during definitive radiotherapy, and (2) correspondingly increase the proportion of patients receiving physician-directed interventions for treatment-related symptoms.

The IMPROVE pilot study will describe the proportion of patients with cancer with changes in physician-perception of treatment-related toxicity that result from routine physician review of PROMs reported during definitive radiotherapy. The IMPROVE study will also describe (1) the proportion of patients with changes in the management of treatment-related symptoms and (2) the type of management changes that result from routine physician review of PROMs reported during definitive radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Able to read and write in English or able to understand/answer questions with the aid of an interpreter
* Histologically confirmed loco-regional to advanced primary cancer, including but not limited to lung cancer, esophageal, or gastro-intestinal cancers at risk of developing radiotherapy-related toxicity.
* Receiving definitive conventionally-fractionated radiation treatment with or without chemotherapy

Exclusion Criteria:

* Patients receiving radiation for palliative intent
* Patients who do not provide informed consent
* Patients who chose to withdraw from the study

Radiation Oncologists

Inclusion criteria:

• Must be the physician overseeing the care of the patient who answers the PROMS

Exclusion criteria:

• Have not provided informed consent

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our study population will be treating radiation oncologists and their primary cancer patients requiring definitive treatment with radiation with or without concurrent chemotherapy as per the inclusion criteria below. Cancer patients receiving stereotactic body radiation therapy or hypo-fractionated definitive radiation will not be recruited as these patients represent a different treatment population with a much lower overall treatment toxicity burden.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranh Voong, MD, Principal Investigator — SKCCC at Johns hopkins
Locations (4):
- United States (4):
  - Bayview Medical Center, Baltimore, Maryland
  - Khinh Voong, Baltimore, Maryland
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 104 patients enrolled in the study. Four patients were excluded from the analysis.
Period: Overall Study
Arm/Group | Patients With Cancer Treated With Definitive-intent Radiotherapy
Started | 104
Completed | 100
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Four patients were excluded from the analysis
Arm/Group | Patients With Cancer Treated With Definitive-intent Radiotherapy
Number analyzed (Participants) | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [61 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian, non-Hispanic | 81
  African American | 13
  Other | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Participants With Change in Their Physician-assessed Burden Score
Description: The primary outcome is patients with any change in physicians-assessed burden scores for at least one radiotherapy on-treatment visit. Lee et al. demonstrated the feasibility of using a global burden score to capture the provider's overall perception of the combined burden of all assessed symptoms, using a visual analogue scale demarcating an aggregate score from 0 to 10. This scale uses anchors at 0, 2, 4, 6, 8, and 10 for no, mild, moderate, severe, life-threatening adverse events, and death, respectively. A 2-point score change correlates to a change to the next anchored score (i.e., mild to moderate, 2 to 4; or moderate to severe, 4 to 6)
Time Frame: Up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cancer Treated With Definitive-intent Radiotherapy
Number analyzed (Participants) | 100
Participants
  Patients with an increased or decreased burden-score of 1 point. | 43
  Patients with an increased or decreased burden-score of ≥ 2 points. | 32
  Patients with no change in burden-score. | 25

2. Secondary Outcome: Participants With Changes in the Management of On-treatment Symptoms
Description: During weekly on-treatment visits and prior to reviewing the patient's PROMs, physicians will formulate an initial symptom management plan based on available clinical data. After reviewing the patient's PROMs, physicians will report participants with changes in recommended interventions due to review of the PROMs.
Time Frame: Up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cancer Treated With Definitive-intent Radiotherapy
Number analyzed (Participants) | 100
Participants
  New Medications/ New Interventions | 29
  Counseling/ Modification of Medications | 39
  Referral to Other Services/ Further Tests | 19

3. Other Pre Specified Outcome: Management Changes as Assessed by a Clinician Feedback Form
Description: At the end of each patient's course of radiotherapy, providers will complete a Clinician Feedback Form that details the types of new management interventions resulting from routine review of the PROMs over the course of definitive radiation.
Time Frame: Up to 2 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 months
Arm/Group | Patients With Cancer Treated With Definitive-intent Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT04589247/Prot_SAP_000.pdf